CLINICAL TRIAL: NCT05241288
Title: Use of ProAir Digihaler in Chronic Obstructive Pulmonary Disease (COPD) - Characterization of Inhalation Metrics From a Cohort of Patient At-risk for Acute Exacerbation of COPD (AECOPD) in an Outpatient Setting
Brief Title: Digihaler in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Wake Forest University Health Sciences (Other); Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-0273
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Results first posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases; Albuterol; Bronchodilator Agents; Respiratory System Agents
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases

STUDY DESIGN:
Intervention Model Description: All participants will receive the intervention consisting of Albuterol eMDPI DS (ProAir® Digihaler®). Participants will be asked to use the ProAir Digihaler as their primary mode of SABA therapy as they would in usual treatment and indicated in the product package insert and Instructions for Use. They will answer a daily self-assessment on the DAQ App, as well as Digihaler metric algorithm-triggered DAQ on the DAQ app. The DAQ will collect yes/no responses to questions focused on change in symptoms. The participants will be contacted once per month to collect COPD Assessment Test (CAT) score and self-reported average albuterol use over the preceding month. They will also be asked about any AECOPD events requiring treatment.
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Albuterol eMDPI DS (ProAir® Digihaler®) (Experimental): This arm will receive the intervention of the Albuterol eMDPI DS for three months.
  Interventions: Combination Product: Albuterol eMDPI DS

INTERVENTIONS:
Combination Product: Albuterol eMDPI DS — Albuterol sulfate electronic multidose dry powder inhaler (Albuterol eMDPI) Digital System (DS) with 3 component devices:
  Device 1: Albuterol eMDPI Device 2: Albuterol eMDPI Patient-facing smart device application (App) Device 3: Digital Health Platform (DHP, Cloud solution)
  Other Names: ProAir® Digihaler®

SUMMARY:
This is a multi-center 3-month study to determine the variation in ProAir Digihaler metrics [peak inspiratory flow (PIF), inhalation volume, number of inhalation events] amongst COPD patients in the ambulatory setting.

DETAILED DESCRIPTION:
The albuterol sulfate electronic multidose dry powder inhaler (Albuterol eMDPI) Digital System (DS) (ProAir® Digihaler®) is the first and only Food and Drug Administration (FDA) approved inhaler rescue medication with a built-in sensor to detect and record inhaler use. The inhaler device measures PIF and the app groups PIF into categories that can help to highlight potential patient inhaler technique errors. This study will deploy this product in COPD patients to establish foundational data on Digihaler metrics in a COPD population at greater risk for COPD exacerbations.

Adult subjects with COPD recruited from two sites [University of North Carolina (UNC) and Wake Forest] will participate in a longitudinal study to collect data regarding the normal variation in Digihaler metrics (PIF, inhalation volume, number of inhalations), a daily self-assessment asking "How are you feeling?" with responses provided on a Likert scale as well as responses to a Digihaler metric algorithm-triggered digital automated questionnaire (DAQ) in a stable COPD population with history of an AECOPD, to assess correlations of Digihaler metrics to daily self-assessment and DAQ responses, correlations of self-reported to actual short acting beta agonist (SABA) use and symptoms, and the changes in inhaler parameters and SABA use around incidental AECOPD.

ELIGIBILITY:
Inclusion Criteria:

* Age >40 years old
* History of cigarette smoking >=10 pack-years
* Established COPD defined as physician diagnosis along with spirometry confirmation [post-bronchodilator (BD) forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC)<0.70] within the last two years and an FEV1 ≤80% predicted
* Regular albuterol use (defined as at least one puff weekly for each of the last four weeks)
* Currently non-hospitalized
* Medical records confirmed history of two moderate AECOPD (defined as use of antibiotic or steroids to treat clinical event consistent with AECOPD) or one severe AECOPD (defined as emergency department/hospital visit) in prior 12 months
* Access to smart phone, tablet or computer and internet
* Willingness to switch current rescue inhaler/device to ProAir Digihaler

Exclusion Criteria:

* Allergy or inability/contraindication to use Albuterol Sulfate
* Any condition that, in the opinion of the site investigator, would compromise the subject's ability to participate in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Drummond, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Albuterol eMDPI DS (ProAir® Digihaler®): This arm will receive the intervention of the Albuterol eMDPI DS for three months.
  Albuterol eMDPI DS: Albuterol sulfate electronic multidose dry powder inhaler (Albuterol eMDPI) Digital System (DS) with 3 component devices:
  Device 1: Albuterol eMDPI Device 2: Albuterol eMDPI Patient-facing smart device application (App) Device 3: Digital Health Platform (DHP, Cloud solution)
Period: Overall Study
Arm/Group | Albuterol eMDPI DS (ProAir® Digihaler®)
Started | 54
Completed | 40
Not Completed | 14

BASELINE CHARACTERISTICS:
Population: Data presented for those participants with both primary and secondary outcome data.
Arm/Group | Albuterol eMDPI DS (ProAir® Digihaler®)
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Mean Variability in Peak Inspiratory Flow (PIF)
Description: PIF is the maximal flow occurring during an inhalation effort, expressed in Liters/minute. Mean and standard deviation of daily PIF measurement collected over three months will be calculated. PIF will be measured using the Digihaler device.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Albuterol eMDPI DS (ProAir® Digihaler®)
Number analyzed (Participants) | 40
Liters/minute | 67.6 (20.3)

2. Primary Outcome: Variability in Peak Inspiratory Flow (PIF) as Measured by Coefficient of Variation
Description: PIF is the maximal flow occurring during an inhalation effort, expressed in Liters/minute. Coefficient of variation (calculated by dividing standard deviation of PIF by the mean of the PIF) of daily PIF measurement collected over three months will be calculated. PIF will be measured using the Digihaler device.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Albuterol eMDPI DS (ProAir® Digihaler®)
Number analyzed (Participants) | 40
Correlation coefficient | 0.286 [0.246 to 0.325]

3. Secondary Outcome: Correlation of Self-Reported Inhaler Use With Actual Inhaler Use
Description: Correlation between self-reported inhaler use and actual inhaler use over three months will be calculated with Spearman rank-order correlation coefficient. Self-reported inhaler use will be determined with an investigator-developed single question categorizing average use over the last four weeks with five groups (not at all, once a week or less, two or three times a week, one or two times a day, three or more times a day). Actual inhaler use will be directly measured via Digihaler device and categorized into one of the five groups described above.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Albuterol eMDPI DS (ProAir® Digihaler®)
Number analyzed (Participants) | 40
Correlation coefficient | -0.385 [-0.413 to -0.357]

4. Secondary Outcome: Mean Variability in Inhalation Volume
Description: Inhalation volume is the volume of air inspired during an inhalation effort, expressed in Liters. The mean and standard deviation of daily inhalation volume measurements collected daily over three months will be calculated. Inhalation volume will be measured using the Digihaler device.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Albuterol eMDPI DS (ProAir® Digihaler®)
Number analyzed (Participants) | 40
Liters | 1.395 (0.598)

5. Secondary Outcome: Variability in Inhalation Volume as Measured by Coefficient of Variation
Description: Inhalation volume is the volume of air inspired during an inhalation effort, expressed in Liters. Coefficient of variation (calculated by dividing standard deviation of inhalation volume by the mean of the inhalation volume) of daily inhalation volume measurement collected over three months will be calculated.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Albuterol eMDPI DS (ProAir® Digihaler®)
Number analyzed (Participants) | 40
Correlation coefficient | 0.426 [0.366 to 0.485]

ADVERSE EVENTS:
Time Frame: From signing of informed consent throughout duration of study, a total of approximately 3 months.
Arm/Group | Albuterol eMDPI DS (ProAir® Digihaler®)
All-Cause Mortality (participants affected / at risk) | 1/54
Serious Adverse Events (participants affected / at risk) | 5/54
Other Adverse Events (participants affected / at risk) | 8/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albuterol eMDPI DS (ProAir® Digihaler®) (N=54)
COPD Exacerbation with hospitalization (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Metastatic Lung Cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Progression of known lung cancer leading to death.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albuterol eMDPI DS (ProAir® Digihaler®) (N=54)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Tremors (Nervous system disorders) | 1 (1)
Oral Candidiasis (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/88/NCT05241288/Prot_SAP_000.pdf